CLINICAL TRIAL: NCT02935374
Title: Effect of Antimicrobial Treatment of Acute Otitis Media on the Intestinal Microbiome in Children: A Randomized Controlled Trial
Brief Title: Effect of Antimicrobial Treatment of Acute Otitis Media on the Intestinal Microbiome in Children
Acronym: AOMMi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OY20167
Record Dates: First submitted 2016-09-28; First posted 2016-10-17 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Acute Otitis Media
Keywords: children; intestinal microbiome; microbiota; antimicrobial course; amoxicillin; amoxicillin-clavulanate; macrolide
MeSH Terms: conditions — Otitis Media | interventions — Amoxicillin; Amoxicillin-Potassium Clavulanate Combination; Macrolides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Amoxicillin (Active Comparator): The children with acute otitis media will be treated with amoxicillin mixture, 100mg/ml, 40mg/kg/d, divided to two daily doses for 7 days.
  Interventions: Drug: Amoxicillin
- Amoxicillin-Potassium Clavulanate (Active Comparator): The children with acute otitis media will be treated with amoxicillin-clavulanate mixture, 80mg/ml, 45mg/kg/d, divided to two daily doses for 7 days.
  Interventions: Drug: Amoxicillin-Potassium Clavulanate
- Wait and see (No Intervention): The children with acute otitis media will be monitored without antimicrobial treatment.
- Macrolide (Other): The children with acute otitis media with known allergy to amoxicillin or amoxicillin-clavulanate will be treated with macrolide and monitored as a separate group, outside randomization.
  Interventions: Drug: Macrolide

INTERVENTIONS:
Drug: Amoxicillin — The children with acute otitis media will be treated with amoxixillin mixture, 100mg/ml, 40mg/kg/d, divided to two daily doses for 7 days.
  Arms: Amoxicillin
Drug: Amoxicillin-Potassium Clavulanate — The children with acute otitis media will be treated with amoxixillin-clavulanate mixture, 80mg/ml, 45mg/kg/d, divided to two daily doses for 7 days.
  Arms: Amoxicillin-Potassium Clavulanate
Drug: Macrolide — The children with acute otitis media with a know allergy to amoxicillin or amoxicillin-clavulanate will be treated with macrolide and monitored separately
  Arms: Macrolide

SUMMARY:
This is a randomized, controlled trial studying the effects of various antimicrobial treatments on the intestinal microbiome of small children. The participating children with acute otitis media are treated wither with amoxicillin, amoxicillin-clavulanate or without antibiotics. The children with allergy to amoxicillin receive a course of macrolide and they will be monitored as a separate group. The main outcomes of this trial are the changes in the intestinal microbiome after the treatment.

DETAILED DESCRIPTION:
Antimicrobial treatment of acute otitis media has been proven efficacious in children. It has been suggested that antimicrobial treatment makes a lot of harm to intestinal microbiome and may thus have effects on the child's health and wellbeing. However, data on these changes and their magnitude is scanty. This is a randomized, controlled trial studying the effects of various antimicrobial treatments on the intestinal microbiome of small children. The participating children with acute otitis media are treated wither with amoxicillin, amoxicillin-clavulanate or without antibiotics. The children with allergy to amoxicillin receive a course of macrolide and they will be monitored as a separate group. The main outcomes of this trial are the changes in the intestinal microbiome after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* acute symptoms of respiratory infection AND
* signs of inflammation on the tympanic membrane in otoscopy AND
* middle ear effusion found in pneumatic otoscopy

Exclusion Criteria:

* Suspected or proven complication of acute otitis media (for example acute mastoiditis or perforated tympanic membrane)
* Severe acute otitis media: severe pain and fever > 39 degrees C
* Bilateral acute otitis media in a child younger than 2 years
* Primary or secondary immunodeficiency or Downs syndrome
* Impaired general condition or suspected severe bacterial infection
* Allergy to both amoxicillin and macrolide
* Acute otorrhea through tympanostomy tube
* Antimicrobial treatment ongoing or during previous 7 days

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2016-11; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Change in the relative abundance of Firmicutes in stool samples | Change from baseline to 10 days
  Change in the relative abundance of Firmicutes in stool samples obtained at baseline and at 10 days after the diagnosis of acute otitis media.

SECONDARY OUTCOMES:
Principal coordinate analysis (PCA) of fecal samples | 10 days
  Principal coordinate analysis (PCA) of the microbiota of fecal samples 10 days after starting treatment to acute otitis media
Change in the relative abundance of Actinobacteria in stool samples | Change from baseline to 10 days
  Change in the relative abundance of Actinobacteria in stool samples obtained at baseline and at 10 days after the diagnosis of acute otitis media.
Change in the relative abundance of Bacteroidetes in stool samples | Change from baseline to 10 days
  Change in the relative abundance of Bacteroidetes in stool samples obtained at baseline and at 10 days after the diagnosis of acute otitis media.
Change in the relative abundance of Proteobacteria in stool samples | Change from baseline to 10 days
  Change in the relative abundance of Proteobacteria in stool samples obtained at baseline and at 10 days after the diagnosis of acute otitis media.
Change in the relative abundance of Verrucomicrobia in stool samples | Change from baseline to 10 days
  Change in the relative abundance of Verrucomicrobia in stool samples obtained at baseline and at 10 days after the diagnosis of acute otitis media.
Change in the relative abundance of Lactobacilli in stool samples | Change from baseline to 10 days
  Change in the relative abundance of Lactobacilli in stool samples obtained at baseline and at 10 days after the diagnosis of acute otitis media.
Change in the relative abundance of Bifidobacteria in stool samples | Change from baseline to 10 days
  Change in the relative abundance of Bifidobacteria in stool samples obtained at baseline and at 10 days after the diagnosis of acute otitis media.
Change in the relative abundance of Faecalibacterium prausnitzii in stool samples | Change from baseline to 10 days
  Change in the relative abundance of Faecalibacterium prausnitzii in stool samples obtained at baseline and at 10 days after the diagnosis of acute otitis media.
Change in the diversity of fecal microbiota measured with the number of operational taxonomic units (OTUs) | Change from baseline to 10 days
  Change in the diversity of fecal microbiota measured with the number of operational taxonomic units (OTUs) from baseline to 10 days after the diagnosis of acute otitis media
Change in the diversity of fecal microbiota measured with Shannon index | Change from baseline to 10 days
  Change in the diversity of fecal microbiota measured with Shannon index from baseline to 10 days after the diagnosis of acute otitis media
Change in the diversity of fecal microbiota measured with Chao index | Change from baseline to 10 days
  Change in the diversity of fecal microbiota measured with Chao index from baseline to 10 days after the diagnosis of acute otitis media
Presence of antimicrobial genes measured with the means of metagenomics | 10 days
  Presence of antimicrobial genes measured with the means of metagenomics at 10 days after the diagnosis of acute otitis media
Proportion of Clostridium difficile -positive fecal samples | 10 days
  Occurrence of Clostridium difficile in fecal samples 10 days after the diagnosis of acute otitis media
Proportion of fecal samples with Extended Spectrum Beta-Lactamase -positive strains | 10 days
  Proportion of fecal samples with Extended Spectrum Beta-Lactamase -positive strains 10 days after the diagnosis of acute otitis media

CONTACTS AND LOCATIONS:
Locations (1):
- Mehiläinen, private practice, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No